CLINICAL TRIAL: NCT04032730
Title: Promoting Engagement in the Drug Resistant TB-HIV Care Continuum in South Africa PRAXIS Study (PRospective Study of Adherence in M/XDR-TB Implementation Science) Aim 2
Brief Title: Promoting Engagement in the Drug Resistant TB-HIV Care Continuum in South Africa PRAXIS Study
Acronym: PRAXIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for the AIDS Programme of Research in South Africa (Network)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Dr Nesri Padayatchi, Deputy Director, Centre for the AIDS Programme of Research in South Africa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CAP 086 AIM 2
Record Dates: First submitted 2018-08-29; First posted 2019-07-25 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Adherence, Patient
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants assigned to the control arm will undergo treatment and care for MDR/XDR-TB as per the South African Department of Health guidelines.
- Intervention (Experimental): Participants assigned to the intervention arm will undergo extensive counselling, participants will be provided with an electronic pillbox that monitors their adherence to one of their TB and one of their ART medication. Based on the recordings provided by the wisepill device we will determine if a participant is adherent to their medication and intervene with counselling, phone calls, home visits and relevant referrals.
  Interventions: Device: Wisepill device

INTERVENTIONS:
Device: Wisepill device — Participants will receive a Wisepill device for TB and ART medications. Participants will receive an exit counselling session prior to being discharged.
  Participants will select the content of a text message to be sent when missing a dose as measured by Wisepill non-opening during medication dose-window.
  Participants will receive a post-discharge phone call by study staff for the purpose of identifying any early challenges or obstacles. All participants may receive a titrated Wisepill intervention (TWI) consisting of a text message, phone call, and/or study home visit triggered by medication non-adherence as detected by Wisepill non-opening.
  All participants will receive a monthly counselling intervention (MCI). Adherence support groups (ASG) will be conducted on a monthly basis.
  Other Names: Adherence Support Groups; Monthly Counselling Intervention; Home Visits; Titrated Wisepill Intervention; Exit Counselling for Discharged patients; Post Discharge Phone Calls
  Arms: Intervention

SUMMARY:
The goal of the proposed study is to enhance adherence and retention in care for M/XDR-TB HIV patients through enhanced standard of care, targeted transition to outpatient medication self-administration prior to hospital discharge, and use of community adherence groups, with an overarching goal of promoting patient engagement in a care continuum.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains the leading cause of morbidity and mortality worldwide among people living with HIV (1). Globally, the incidence of multidrug-resistant tuberculosis (MDR-TB) and extensively drug resistant tuberculosis (XDR-TB), the most drug-resistant forms of TB, has approximately doubled over the past fifteen years (1-3). Nowhere has this increased incidence generated more concern than in South Africa where interactions between TB and generalized HIV epidemics are causing 'explosive' TB incidence (4-6) and case-fatality are threatening to undermine the progress reached with antiretroviral therapy (ART) (7, 8).

Medication adherence, a key predictor of outcomes in M/XDR-TB and HIV treatment, is understudied in high burden TB-HIV settings (9-11). Patient losses during transitions in the care continuum are frequent (12), increase mortality and limit control of the linked epidemics. Demands of M/XDR-TB HIV treatment are severe including extraordinary pill burden, severe adverse effects, lengthy treatment, isolation and stigma with few parallels in modern medicine (13-15).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. MTB culture positive with at least isoniazid and rifampicin resistance OR Molecular drug susceptibility test confirming resistance to at least isoniazid and rifampicin OR Polymerase chain reaction test (Xpert MTB/RIF) result showing MTB positive and RIF resistance. OR MTB positive with Rifampicin monoresistance
3. Initiating treatment for M/XDR-TB which includes Bedaquiline (BDQ) or Moxifloxacin/Levaquin
4. Have capacity for informed consent
5. HIV Positive Patients: on ART or initiating ART within the following 4 weeks as per clinician recommendation

Exclusion Criteria:

1. Pregnancy
2. Prisoners
3. Discretion of IOR or clinician

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2018-04-29 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Adherence in M/XDR-TB HIV outcomes | 9-24 months
  The number of participants that are adherent to their TB and ARV medication as assessed by:
  * the use of wisepill device (electronic pill box). 2 wisepill devices are provided to participants in the intervention arm, one for their ART medication and one for their TB medication (namely Bedaquiline).
  * By self reporting via 7-day recall and 30-day recall
  * By self reporting via Visual analogue scale
Retention in care | 9-24 months
  Retention in care will be assessed by loss to follow-up.
TB treatment outcomes | 9-24 months
  The number of participants with TB treatment outcomes as assessed by death or culture conversion.

CONTACTS AND LOCATIONS:
Overall Officials: Nesri Padayatchi, Principal Investigator — Deputy Director
Locations (1):
- King Dinuzulu Hospital, Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: Undecided